CLINICAL TRIAL: NCT05259384
Title: Comparison Between Robotic and Laparoscopic Surgery for Patients With Pancreatic Cystic Neoplasms
Brief Title: Robotic Versus Laparoscopic Surgery for Patients With Pancreatic Cystic Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daimh-ROBOTIC-PCN
Record Dates: First submitted 2021-04-21; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The enrolled candidates will be split into two subgroups(PD group or DP group) based on the location of their neoplasms. Every subgroups will be divided into two parallel groups by the randomization of intervention plan(lap surgery or robotic surgery)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MIPD-ROB (Experimental): Patients with PCN locates HEAD and NECK of pancreas who were randomized to ROBOTIC pancreaticoduodenectomy.
  Interventions: Procedure: Robotic pancreaticoduodenectomy
- MIPD-LAP (Active Comparator): Patients with PCN locates HEAD and NECK of pancreas who were randomized to LAPAROSCOPIC pancreaticoduodenectomy.
  Interventions: Procedure: Laparoscopic pancreaticoduodenectomy
- MIDP-ROB (Experimental): Patients with PCN locates BODY and TAIL of pancreas who were randomized to ROBOTIC distal pancreatectomy.
  Interventions: Procedure: Robotic Distal Pancreatectomy
- MIDP-LAP (Active Comparator): Patients with PCN locates BODY and TAIL of pancreas who were randomized to LAPAROSCOPIC distal pancreatectomy.
  Interventions: Procedure: Laparoscopic Distal Pancreatectomy

INTERVENTIONS:
Procedure: Robotic pancreaticoduodenectomy — The Intervention of MIPD-ROB group
  Arms: MIPD-ROB
Procedure: Laparoscopic pancreaticoduodenectomy — The Intervention of MIPD-LAP group
  Arms: MIPD-LAP
Procedure: Robotic Distal Pancreatectomy — The Intervention of MIDP-ROB group
  Arms: MIDP-ROB
Procedure: Laparoscopic Distal Pancreatectomy — The Intervention of MIDP-LAP group
  Arms: MIDP-LAP

SUMMARY:
Pancreatic cystic neoplasm (PCN) is a type of neoplastic lesion formed by the proliferation of pancreatic duct or acinar epithelial cells and retention of pancreatic secretions. The tumor can be located in the head and neck of the pancreas or the body and tail of the pancreas. Conventionally, open pancreaticoduodenectomy or open distal pancreatectomy was performed for patients with PCN locates either at the head or tail. In the ear of minimally invasive pancreatic surgery, when compared with open surgery, laparoscopic technology or Da Vinci robotic technology can avoid some open procedures limitations.

Here we design this prospective randomized clinical trial to compare robotic surgery to laparoscopic surgery for the treatment of PCN and verify the safety and feasibility of both two minimally invasive procedures.

DETAILED DESCRIPTION:
Background: Pancreatic cystic neoplasm (PCN) is a type of neoplastic lesion formed by the proliferation of pancreatic duct or acinar epithelial cells and retention of pancreatic secretions. Its heterogeneity is large, which can be benign, borderline, and poor differentiation and even evolve into pancreatic cancer. The tumor can be located in the head and neck of the pancreas or the body and tail of the pancreas. Some patients may be accompanied by recurrent pancreatitis, abdominal pain, nausea, vomiting, jaundice, and other gastrointestinal symptoms, usually with the help of abdominal ultrasound and endoscopy, ERCP, CT, nuclear magnetic, or MRCP imaging The examination can diagnose the disease. For PCN patients with large tumors, risk of malignant transformation, and accompanying symptoms that affect the quality of life, surgery is an effective treatment.

Based on the conventional routine treatment, open pancreaticoduodenectomy or open distal pancreatectomy was performed for patients with PCN locates either at the head or tail.

After more than 20 years of development, minimally invasive pancreatic surgery technology can be divided into two categories: laparoscopic technology and Da Vinci robotic technology. In general, compared with open surgery, minimally invasive pancreatic surgery technology can avoid some open procedures limitations, reduce the loss of intraoperative body fluid and its impact on the internal environment, and avoid excessive disturbance to other abdominal organs. It also helps reduce the pain of patients and shorten the length of hospital stay. Because most PCNs are benign or borderline tumors, such patients are eligible for minimally invasive pancreatic surgery.

Aim and Hypothesis: Here we design this prospective randomized clinical trial to compare robotic surgery to laparoscopic surgery for the treatment of PCN and verify the safety and feasibility of both two minimally invasive procedures. We conduct a single-center prospective randomized clinical trial to compare the outcomes of different minimally invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older;
2. Diagnosed as PCN;
3. Patients with head or neck PCNs are eligible for minimal invasive PD, or patients with distal PCNs are eligible for minimal invasive DP.

Exclusion Criteria:

1. Not a PCN base on the sample's pathology;
2. Procedure change from MIDP/MIPD to others during the operation;
3. ASA more than 4;
4. Patients or families deny certain treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-17 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Complication Rate | up to 90 days
  The rate of frequency of Clavein-Dindo Grade II-IV complication

SECONDARY OUTCOMES:
Postoperative length of stay | during the treatment
  The mean of postoperative length of stay
VAS score | up to 90 days
  patients complain of pain after surgery, 0-10, 10 means the greatest pain
Grade B and C pancreatic fistula | up to 90 days
  The frequency of grade B or C pancreatic fistula
QOL score | up to 90 days
  Quality of life after surgery, greater means higher life satisfaction
Expense | during the treatment
  The amount of treatment expense and certain procedure expense
90-day death rate | up to 90 days
  The rate of death within 90 days after surgery
The rate of spleen-preservation | up to 90 days
  For DP groups, the rate of spleen being preserved

CONTACTS AND LOCATIONS:
Overall Officials: MENGHUA Dai, M.D., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: No